CLINICAL TRIAL: NCT06936241
Title: Effect of Circuit Weight Training on Functional Capacity and Quality of Life in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alhasnaa Sayed Farouk Helal, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005445
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circuit weight training and traditional physical therapy program (Experimental): The participants will do Circuit Weight Training in addition to traditional physical therapy program for 8 weeks
  Interventions: Other: Circuit weight training; Other: Traditional physical therapy program
- Traditional physical therapy program (Active Comparator): The participants will receive traditional physical therapy program only for 8 weeks
  Interventions: Other: Traditional physical therapy program

INTERVENTIONS:
Other: Circuit weight training — The Circuit Training protocol will be performed as follows:
  wall push-up, bridge on floor, single leg bridge, bird dog, windshield wiper, march in place, ball squat, squat with an overhead press, reverse pendulum, jumping rope, and spinal twist, 30-35 minutes, 3 times a week for 8 weeks
  Arms: Circuit weight training and traditional physical therapy program
Other: Traditional physical therapy program — The participants will receive traditional physical therapy program in the form of therapeutic exercises to keep daily living activity by restoring the strength of flexors and abductors of the shoulder joint using the shoulder wheel and ladder. It will be performed 3 times per week for eight weeks

SUMMARY:
The study is aimed at studying the effects of Circuit Weight Training (CWT) on functional capacity and quality of life in breast cancer patients.

DETAILED DESCRIPTION:
Breast Cancer is the most common cancer among women in Egypt causing 22 percent of all cancer-related female deaths. It is the most commonly diagnosed cancer, accounting for nearly a quarter of all cancer cases globally.

With improvements in early detection, surgery, and adjuvant therapy for breast cancer, long-term survival and cure are becoming possible. Despite providing longer survival with early diagnosis of breast cancer, the treatment leaves sequelae with adverse effects such as influence on functional capacity, fatigue, depression, neuropathic lymphoedema, low immunity, and loss of flexibility. All of these effects end up affecting the quality of life (QoL), Imbalance, gait dysfunction, and falls may have particularly severe consequences in breast cancer survivors due to comorbidities increasing the risk of fall-related injury, secondary decline in physical activity, and subsequent functional decline.

Given the profound effects that imbalance, gait dysfunction, and falls have on functional independence, QOL, and long-term health and survivorship, the treatment or prevention of these symptoms is an essential component of cancer rehabilitation for all survivors.

Furthermore, the need for this study is developed from the lack of quantitative knowledge and information in the published studies about the effect of Circuit Weight Training (CWT) on functional capacity and quality of life in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female with age between 35-45.
* Body Mass Index (BMI) < 25.
* Patients diagnosed with non-metastatic (Stage 0-III) breast cancer.
* All patients who are treated by neoadjuvant chemotherapy before surgery.

Exclusion Criteria:

* Patients diagnosed with cancer metastasis.
* Patients diagnosed with diseases of the nervous system (Parkinson's disease, peripheral nerve palsy) skeletal system (inflammatory diseases, scoliosis >10 Cobb angle), or rheumatic diseases.
* Patients with any current visual impairment that affected their daily living, vestibular disorder, neurological disorder, cognitive disorder, and any further medical condition that would prohibit them from participating safely.

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of quality of life | 8 weeks
  The 12-Item Short Form Survey (SF-12) is the abridged practical form of the SF-36. It is a widely used screening device for measuring physical, mental, and social well-being to assess quality of life. it consists of 2 components: Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12). Its score ranges between 0-100. Higher score indicates better health.
Assessment of functional capacity | 8 weeks
  The 2-minute step test (TMST) will be used to measure exercise capacity for all participants in the study before and after treatment.
  The test simply requires that participants march in place as fast as possible for 2 minutes while lifting the knees to a height midway between their patella and iliac crest when standing. Performance on the test is defined as the number of right-side steps of the criterion height completed in 2 minutes.

SECONDARY OUTCOMES:
Postural stability test | 8 weeks
  It will be used to measure static balance by measuring posture sway by using the Biodex balance system. the overall stability index will be measured; lower score of overall stability index indicates better balance.
Limits of stability test | 8 weeks
  t will be used to measure dynamic balance by using the Biodex balance system. Higher directional control and excursion scores with lower reaction time indicate better voluntary balance control.
Single leg stability test | 8 weeks
  It will be used to assess unilateral balance with progressive instability. Lower stability indexes represent better single-leg balance and neuromuscular control.
Assessment of muscle strength | 8 weeks
  A hand-held dynamometer will be used to assess muscular strength of specific muscles of upper and lower limbs by quantifying the maximum force exerted during specific movement, with higher values indicating greater strength.

CONTACTS AND LOCATIONS:
Overall Officials: Maher H Ibrahim, Professor, Study Director — Cairo University; Heba A. Abdulghafar, Professor, Study Chair — Cairo University
Locations (1):
- Alhasnaa Sayed Farouk, Giza, Egypt